CLINICAL TRIAL: NCT05714631
Title: A Single-blind Randomized Placebo Controlled Trial of Lidocaine Patches for Opioid Reduction in Geriatric Rib Fracture Patients Admitted to the Hospital
Brief Title: Lidocaine Patches in Elderly Patients With Traumatic Rib Fractures
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor Enrollment
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Jacob Peschman, MD, Assistant professor of surgery, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO44982
Record Dates: First submitted 2023-01-26; First posted 2023-02-06 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Rib Fractures
MeSH Terms: conditions — Rib Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Standard of care group (No Intervention): Patients in the standard of care will not be receiving any lidocaine or placebo patches. The aim of this group is to control for the placebo effect
- Placebo group (Placebo Comparator)
  Interventions: Other: Placebo Patch
- Intervention group (Experimental)
  Interventions: Drug: 4% Lidocaine Patch

INTERVENTIONS:
Other: Placebo Patch — Transdermal placebo patch
  Arms: Placebo group
Drug: 4% Lidocaine Patch — Transdermal patch
  Arms: Intervention group

SUMMARY:
Many patients are prescribed lidocaine patches for rib fractures despite mixed evidence to their efficacy. The outcome of this trial offers significant benefit to patient care if it finds benefit of their use or if it does not. Reducing opioid use and increasing functional outcomes in geriatric patient suffering rib fractures can improve quality of life and ability to return to prior levels of function. Limiting the need for opioid prescriptions dispensed in the community, particularly to vulnerable geriatric individuals, is also a key aspect in curbing the opioid epidemic. However, even if no difference is found, it would support stopping the use of lidocaine patches in this population as a waste of money and resources. The novel approach of adding the 3rd arm to assess for placebo effect will also carry clinical value, as a placebo effect that reduces opioid use may in fact be enough to support continued use of the products given their overall low side effect risk profile compared to opioids and other pain control medications.

DETAILED DESCRIPTION:
Many patients are prescribed lidocaine patches for rib fractures despite mixed evidence to their efficacy. The outcome of this trial offers significant benefit to patient care if it finds benefit of their use or if it does not. Reducing opioid use and increasing functional outcomes in geriatric patient suffering rib fractures can improve quality of life and ability to return to prior levels of function. Limiting the need for opioid prescriptions dispensed in the community, particularly to vulnerable geriatric individuals, is also a key aspect in curbing the opioid epidemic. However, even if no difference is found, it would support stopping the use of lidocaine patches in this population as a waste of money and resources. The novel approach of adding the 3rd arm to assess for placebo effect will also carry clinical value, as a placebo effect that reduces opioid use may in fact be enough to support continued use of the products given their overall low side effect risk profile compared to opioids and other pain control medications

AIM 1: Determine if a 3-armed placebo controlled randomized trial evaluating the efficacy of 4% lidocaine patches is feasible on a large scale with up to 500 enrolled patients across multiple institutions.

Objective 1: Evaluate the study design, randomization system, drug delivery and placebo creation processes to determine barriers to a larger multicenter study design.

AIM 2: Determine if the use of 4% lidocaine patches decreases the utilization of opioids in geriatric (Age ≥65) patient with rib fractures and minimal other injuries by 50% or more during the first 72 hours of hospitalization.

Objective 2: Determine an appropriate target opioid reduction rate and appropriate enrollment numbers for a future a larger scale trial. We suspect a 50% opioid reduction may be larger than would be expected for a single aspect of multimodal pain control treatment. While the study will be powered to identify this difference, it is more likely that a 20-40% reduction could be achieved and therefore help determine appropriate power calculations for a future trial.

AIM 3: Determine if there is a potential placebo effect of topical patch therapy.

Objective 3: Utilizing a 3rd arm increases the number of patients needed to enroll but will help clarify if there is a significant placebo effect from the application of a non-medicated patch over rib fractures. There may be clinical benefit from this placebo effect itself which would need to be accounted for clinical recommendations generated from this and future studies.

AIM 4: Include post discharge opioid usage in analysis to determine the prolonged pain needs of patients suffering rib fractures.

Objective 4: Assess the feasibility of incorporating opioid prescription data using the Wisconsin Prescription Drug Monitoring Program (WI PDMP)as part of a clinical trial as a measure of post discharge opioid use.

Approved study staff will be screening the trauma surgery patients list. Elderly patients (>/=65) with traumatic rib fractures will be approached within 24 hours after admission. Approved study staff will explain the project and informed consent in its entirety. Patients will then be randomized to one of 3 arms: 4% Lidocaine Patches, Placebo, Standard of Care (no lidocaine patch). Randomization will take place using RedCap database. The patients will receive the study drug or placebo as recommended by the manufacturer as 12 hours on, 12 hours off regimen. The patch location will be selected by the patient and nurse based on site of maximal pain. The patient will receive 1 drug or placebo patch for 1-3 rib fractures, 2 patches if 4-6 rib fractures, and 3 patches (maximum dose) if & or more fractures. The 4% Lidocaine patches will be obtained from the Froedtert Investigational Drug Office and dispensed with enough supply to last for 3 patch cycles in 5 days. The patches will then have kinesio tape (designed for topical application) applied over the patch to blind the patients to whether it is a study drug or placebo. For placebo, a double thickness similarly shaped piece of kinesio tape will be used. Based on drug efficacy, all patches can be prepared at the time of study enrollment and remain viable for use during the duration of the study. Patients in the standard of care arm will not receive a patch. All other pain medications will be prescribed at the discretion of treating providers based on standard of care (see section 52.1 Pain Management Protocol Lidocaine RCT). Approved study staff will be accessing patient's electronic medical record 5 days after enrollment; approved study staff will gather information regarding pain score (scored out of 10) and oral morphine equivalent (OME). Dr. Jacob Peschman is the director of outpatient services; he will be accessing patient's 30-day post discharge opioid use utilizing the Wisconsin Prescription Drug Monitoring Program (PDMP). Patients will be approached by approved study staff 30-days post discharge. Patients will be asked several questions regarding pain score and control.

ELIGIBILITY:
Inclusion Criteria:

* age>/= 65 years
* Patients with injuries meeting an AIS score </=2
* Patients admitted to trauma service
* Patients able to consent

Exclusion Criteria:

* Age <65 years
* Unable to consent
* Chronic pain medication usage; defined as >/= 3 weeks of >/= 30 mg oral morphine equivalent
* History of allergic reaction to lidocaine or adhesive tape
* Prisoners
* Patient will be excluded if pain is worse in non-ribs location
* Patient will be excluded if he has injuries not meeting our criteria

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Oral Morphine equivalent | Up to 30-days. From date of randomization until the date of patient discharge
Patient reported pain score (scale from 0-10) | Up to 30-days. From date of randomization until the date of patient discharge

SECONDARY OUTCOMES:
30-day opioid usage | 30-day post discharge using the Wisconsin Prescription Drug Monitoring Program

CONTACTS AND LOCATIONS:
Locations (1):
- Abdul Hafiz Al Tannir, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No